CLINICAL TRIAL: NCT02418013
Title: A Randomized, Double-blinded and Placebo-controlled Pilot Clinical Trial to Evaluate the Potential Efficacy and Safety of Human Umbilical Cord Blood and Plasma by Clinical Markers of Frailty in Adult Who Defined Pre-Frailty
Brief Title: Clinical Trial to Evaluate the Potential Efficacy and Safety of Human Umbilical Cord Blood and Plasma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, Myung Ryool Park, Professor, Bundang CHA Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHAIRB_BD_V.5.1_F011
Record Dates: First submitted 2015-03-26; First posted 2015-04-16 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Aging
Keywords: Frailty; Umbilical cord blood; Plasma; Randomized trial; Double-blinded trial; Placebo-controlled trial
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fresh cord blood(experimental group A) (Experimental): 16 males and 16 females are assigned to the experimental group A. Dropout is 20 percent in each gender.
  Interventions: Other: Fresh cord blood(experimental group A)
- Frozen cord blood(experimental group B) (Experimental): 16 males and 16 females are assigned to the experimental group B. Dropout is 20 percent in each gender.
  Interventions: Other: Frozen cord blood(experimental group B)
- Frozen plasma(experimental group C) (Experimental): 16 males and 16 females are assigned to the experimental group C. Dropout is 20 percent in each gender.
  Interventions: Other: Frozen plasma(experimental group C)
- Placebo group (Placebo Comparator): 16 males and 16 females are assigned to the Placebo group. Dropout is 20 percent in each gender. Total participants are 64 in males and 64 in females.
  Interventions: Other: Placebo group

INTERVENTIONS:
Other: Fresh cord blood(experimental group A) — 1. Cord blood is administered through intravenous at CHA clinical trail institute.
  2. Chlorpheniramine maleate at the concentration of 0.6ml/10kg is administered prior to the treatment.
  Arms: Fresh cord blood(experimental group A)
Other: Frozen cord blood(experimental group B) — 1. Cord blood is administered through intravenous at CHA clinical trail institute.
  2. Chlorpheniramine maleate at the concentration of 0.6ml/10kg is administered
  Arms: Frozen cord blood(experimental group B)
Other: Frozen plasma(experimental group C) — 1. Cord blood is administered through intravenous at CHA clinical trail institute.
  2. Chlorpheniramine maleate at the concentration of 0.6ml/10kg is administered
  Arms: Frozen plasma(experimental group C)
Other: Placebo group — A placebo agent is administered through intravenous at CHA clinical trail institute.
  It should be certain that when administered, participants are not aware of which treatments are preformed.
  Arms: Placebo group

SUMMARY:
This study aims to carry out a safety evaluation of human cord blood and frozen plasma as treatment for pre-frailty , to assess whether the treatment can prevent and improve the aging process, and to identify useful clinical markers of frailty.

The study is a randomized, double-blinded and placebo-controlled pilot clinical Trial conducted at CHA clinical trial institute.

DETAILED DESCRIPTION:
Assessment criteria for the study include (1) clinical indicators-weight loss, a decrease in physical activity, weak grip strength, depression; (2) Short Physical Performance Battery(SPPB); (3) SF-36; (4)cardiac output; (4)biomarkers for oxidative stress, inflammation and immune response; (5) methylation; (6) mitochondria DNA copy number; (7) growth factors; (8) antioxidant capacity; (9) hormone assay; (10) genome assay; (11) metabolite; (12) safety of intravenous administration.

Participants will be randomly assigned to three experimental groups and one control group in a ratio of 1:1:1:1. At second visit, the participants will be administered with experimental and placebo agents. Follow-up visits are expected to be at 7 days, 1 and 6 months after the first treatment. Sixth visit is the completion of it.

Primary end points are defined as severe clinical abnormalities, which could be observed until 1 month after administration of blood-derived products, including death, pulmonary embolism, stroke, respiratory stress and hospitalization due to abnormal findings in laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of pre-frailty
2. One or two scores in Simple FRAIL questionnaire
3. Aged 55 or over
4. Willing and able to be hospitalized according to the research plan
5. Able to participate in our research during 12 months
6. For women, they must be diagnosed with menopause or infertility

Exclusion Criteria:

1. Diagnosis of being irreversible disabled
2. Dementia or cognitive impairment clinically relevant to it
3. Unable to perform tasks required for analysis of primary end point
4. Scheduled to receive organ transplantation
5. Hemoglobin < 8 g/dl; white blood cells count <3000/mm3; absolute Neutrophil count < 500/dl; Thrombocyte count <80,000/mm3; , AST/ALT or ALP > 3 times the normal level
6. Hemoglobin >17g/dl for male and >16 g/dl for female
7. Diagnosis of cancer within 5 years or having the possibility to contract cancer
8. Anticancer chemotherapy and radiation therapy
9. History (within 6 months) of acute diseases such as myocardial infarction, unstable angina, stroke, bone fracture
10. Hormone therapy within 6 months
11. Recent and current use of Immunosuppressive drug or HIV patients
12. History of hospitalization due to infectious disease such as pneumonia within one year
13. Previous (within one months) or current participants in other clinical trials
14. Severe kidney (eGFR< 30) and heart failure (Class III/IV)
15. Any participants who, in the opinion of the investigators, are considered to have safety problems and/or not to perform tasks successfully
16. History of drug or alcohol abuse
17. Chronic Hepatitis B or C: history taking
18. Known or suspected pregnancy (Women must be subjected to pregnancy test)
19. Hypersensitive to dimethyl sulfoxide(DMSO)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Changes in scores of Short Physical Performance Battery (SPPB) as a measure of efficacy for anti-aging effects | 7 days after transplantation
  The investigators will assess changes in scores from baseline at 7 days after transplantation. After normality test, either unpaired t-test or wilcoxon rank sum test will be conducted.

SECONDARY OUTCOMES:
Hand grip strength (in kg) as a measure of efficacy for anti-aging effects | 6 months period after transplantation
  The test is scheduled to be conducted at the day of transplantation and at 1 week , 1 month, 6 months after the treatments. After normality test on the average difference, either unpaired t-test or wilcoxon rank sum test will be conducted for statistical analysis.
  The followings are diagnosis criteria for frailty based on hand grip strength(in kg):
  Male
  1. equal or less than 18 kg for the participants with BMI (body mass index)≤21.89
  2. equal or less than 23 kg for the participants with 22.02 <BMI≤23.63
  3. equal or less than 21.5 kg for the participants with 23.67<BMI≤24.63
  4. equal or less than 25 kg for the participants with BMI>24.88
  Female
  1. equal or less than 12.2 kg for the participants with BMI (body mass index)≤22.52
  2. equal or less than 13 kg for the participants with 22.53<BMI ≤24.23
  3. equal or less than 14.5 kg for the participants with 24.24<BMI ≤26.44
  4. equal or less than 13 k
SF_36(The Short Form (36) Health Survey) as a measure of improvement in the quality of life | 6 months period after transplantation
  The test is scheduled to be conducted at the day of transplantation (2nd visit) and at 1 week (3rd visit), 1 month (4th visit), 6 months (5th visit) after the treatments. The investigators will assess changes compared to baseline which will be measured at the day of transplantation. After normality test on the average difference, either unpaired t-test or wilcoxon rank sum test will be conducted for statistical analysis.
Biomarkers for oxidative stress and inflammation as a measure of efficacy for anti-aging effects | 6 months period after transplantation
  The test is scheduled to be conducted at the day of transplantation (2nd visit) and at 1 week (3rd visit), 1 month (4th visit), 6 months (5th visit) after the treatments. Changes in biomarkers such as CRP, IL-1,6, IL-10, LIF, D-dimer, fibrinogen, TNF-α, CBC with differential, malondialdehyde, 4-hydroxynonenal will be assessed. After normality test on the average difference, either unpaired t-test or wilcoxon rank sum test will be conducted for statistical analysis.
Biomarkers for immune response as a measure of efficacy for anti-aging effects | 6 months period after transplantation
  The test is scheduled to be conducted at the day of transplantation (2nd visit) and at 1 week (3rd visit), 1 month (4th visit), 6 months (5th visit) after the treatments. The investigators will assess changes of the immune-related biomarkers compared to baseline which will be measured at the day of transplantation. After normality test on the average difference, either unpaired t-test or wilcoxon rank sum test will be conducted for statistical analysis.
  Followings are immune markers to be tested
  -Eotaxin, FGF-2,Flt-3 Ligand ,Fractalkine,G-CSF, GM-CSF, GRO, IFNa2, IFNr, IL-1a, IL-1b, IL-1ra, IL-2, IL-3, IL-4 ,IL-5 ,IL-6 ,IL-7, IL-8, IL-9, IL-10, IL-12(p40), IL-12(p70), IL-13, IL-15, IL-17, IP-10, MCP-1, MCP-3, MDC, MIP-1a, MIP-1b, PDGF-AA, PDGF-AB/BB, RANTES, sCD40L, sIL-2Ra TGFa, TNFa,TNFb, VEGF
Adrenal cortical hormone levels as a measure of efficacy for anti-aging effects | Up to 6 months after transplantation
  The test is scheduled to be conducted at the day of transplantation (2nd visit) and at 1 week (3rd visit), 1 month (4th visit), 6 months (5th visit) after the treatments. The investigators will assess changes in hormone levels compared to baseline which will be measured at the day of transplantation.
  After normality test on the average difference, either unpaired t-test or wilcoxon rank sum test will be conducted for statistical analysis.
Telomere length as a measure of efficacy for anti-aging effects | 6 months period after transplantation
  The test is scheduled to be conducted at the day of transplantation (2nd visit) and at 1 week (3rd visit), 1 month (4th visit), 6 months (5th visit) after the treatments. Whether the treatments protect telomere from shortening will be investigated through the comparison analysis.
  After normality test on the average difference, either unpaired t-test or wilcoxon rank sum test will be conducted for statistical analysis.
Body composition as a measure of efficacy for anti-aging effects | 6 months period after transplantation
  The test is scheduled to be conducted at the day of transplantation (2nd visit) and at 1 week (3rd visit), 1 month (4th visit), 6 months (5th visit) after the treatments. The investigators will assess changes of body composition compared to baseline which will be measured at the day of transplantation.
  After normality test on the average difference, either unpaired t-test or wilcoxon rank sum test will be conducted for statistical analysis.
Aging-related genetic and epigenetic markers as a measure of efficacy for anti-aging effects | 6 months period after transplantation
  The test is scheduled to be conducted at the day of transplantation (2nd visit) and at 1 week (3rd visit), 1 month (4th visit), 6 months (5th visit) after the treatments. The investigators will assess changes of aging-related genetic markes (e.g ELOVL2. ) compared to baseline which will be measured at the day of transplantation.
  After normality test on the average difference, either unpaired t-test or wilcoxon rank sum test will be conducted for statistical analysis.
mitochondria DNA copy number as a measure of efficacy for anti-aging effects | 6 months period after transplantation
  The test is scheduled to be conducted at the day of transplantation (2nd visit) and at 1 week (3rd visit), 1 month (4th visit), 6 months (5th visit) after the treatments. Mitochondria DNA copy number of participants will be compared among the treatment groups.
  After normality test on the average difference, either unpaired t-test or wilcoxon rank sum test will be conducted for statistical analysis.
Aging-related growth factors(GDF11, GDF15, Myostatin) as a measure of efficacy for anti-aging effects | 6 months period after transplantation
  The test is scheduled to be conducted at the day of transplantation (2nd visit) and at 1 week (3rd visit), 1 month (4th visit), 6 months (5th visit) after the treatments. The investigators will assess changes compared to baseline which will be measured at the day of transplantation. The factors will be compared among the treatment groups. After normality test on the average difference, either unpaired t-test or wilcoxon rank sum test will be conducted for statistical analysis.
DNA damage extent (8-hydroxyguanine level) as a measure of efficacy for anti-aging effects | 6 months period after transplantation
  The test is scheduled to be conducted at the day of transplantation (2nd visit) and at 1 week (3rd visit), 1 month (4th visit), 6 months (5th visit) after the treatments. The investigators will assess changes of 8-hydroxyguanine in white blood compared to baseline which will be measured at the day of transplantation.
  After normality test on the average difference, either unpaired t-test or wilcoxon rank sum test will be conducted for statistical analysis.
Changes in scores of Short Physical Performance Battery (SPPB) as a measure of efficacy for anti-aging effects | 6 months period after transplantation
  The test is scheduled to be conducted at the day of transplantation (2nd visit) and at 1 week (3rd visit), 1 month (4th visit), 6 months (5th visit) after the treatments.
  The investigators will assess changes in scores compared to baseline which will be measured at the day of transplantation.
  After normality test on the average difference, either unpaired t-test or wilcoxon rank sum test will be conducted for statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Myung Ryool Park, PhD, Principal Investigator — orthopedics
Locations (1):
- Bundang CHA hospital, Seongnam, Bundanggu, South Korea